CLINICAL TRIAL: NCT05110950
Title: Diagnostic Accuracy of Endobronchial Ultrasound Needle Aspiration With and Without Suction: a Single-center Randomized Controlled Trial
Brief Title: Endobronchial Ultrasound Needle Aspiration With and Without Suction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Stefano Gasparini, Professor, Università Politecnica delle Marche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: AspiraTE2021
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Mediastinal Lymphadenopathy; Hilar Lymphadenopathy; Lymphoma; Lung Neoplasms; Sarcoidosis; Tuberculosis; EGF-R Positive Non-Small Cell Lung Cancer; PDL1 Gene Mutation; ALK Translocation; ROS1 Gene Mutation
MeSH Terms: conditions — Lymphoma; Lung Neoplasms; Sarcoidosis; Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the pathologist and the patient are not aware of the type of adopted aspiration technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No suction EBUS-TBNA (Active Comparator): In this technique the stylet is slowly removed without any kind of device in order to avoid active suction.
  Interventions: Procedure: No suction EBUS-TBNA
- Passive suction through dedicated EBUS-TBNA syringe (Active Comparator): After rapid stylet removal, suction is applied through a vacuteiner syringe, without active aspiration.
  Interventions: Procedure: Passive suction through dedicated EBUS-TBNA syringe
- Manual applied suction EBUS-TBNA through a pistol-grip syringe holder (Active Comparator): After rapid stylet removal, suction is applied through Cameco syringe pistol, that can apply active suction manually.
  Interventions: Procedure: Manual applied suction EBUS-TBNA through a pistol-grip syringe holder

INTERVENTIONS:
Procedure: No suction EBUS-TBNA — The needle is moved from a side to side of the lymphnode for 15 times. Each lymphnode is sampled three times.
  The samples obtained will be examined on-site by experienced blinded cytopathologist.All specimens obtained will be send to definitive cytological and histological evaluation and the final diagnosis will be collected and reported on CRFs.
  Arms: No suction EBUS-TBNA
Procedure: Passive suction through dedicated EBUS-TBNA syringe — The needle is moved from a side to side of the lymphnode for 15 times. Each lymphnode is sampled three times.
  The samples obtained will be examined on-site by experienced blinded cytopathologist.All specimens obtained will be send to definitive cytological and histological evaluation and the final diagnosis will be collected and reported on CRFs.
  Arms: Passive suction through dedicated EBUS-TBNA syringe
Procedure: Manual applied suction EBUS-TBNA through a pistol-grip syringe holder — The needle is moved from a side to side of the lymphnode for 15 times. Each lymphnode is sampled three times.
  The samples obtained will be examined on-site by experienced blinded cytopathologist.All specimens obtained will be send to definitive cytological and histological evaluation and the final diagnosis will be collected and reported on CRFs..
  Arms: Manual applied suction EBUS-TBNA through a pistol-grip syringe holder

SUMMARY:
The main purpose of the present study is to compare the diagnostic yield of different aspiration techniques in Ultrasound-guided Transbronchial Needle Aspiration (EBUS-TBNA) in the diagnosis of hilar/mediastinal adenopathy

DETAILED DESCRIPTION:
The role of ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) for the diagnosis of hilar/mediastinal adenopathy is well established. However, different aspiration techniques are available and it's not clear if there's a significant difference between suction vs no suction aspiration. Of great interest is the role of different aspiration techniques in EBUS-TBNA in determining the diagnostic yield for histopathological evaluation, including molecular biology and PD-L1 amplification assessment in lung cancer diagnosis.

In this context, no comparative studies between suction and no suction aspiration have been performed; moreover, considering only suction techniques, no studies evaluated if there's a difference between aspiration with EBUS dedicated syringe and manual aspiration through Cameco syringe. It is very important for clinical practice to definitively assess the non inferiority of no suction techniques in EBUS-TBNA in terms of diagnostic yield, and to provide information regarding the quality of histologic sample to define the best diagnostic strategy.

The study is focused on a minimum of 306 patients who have at least one hilar/mediastinal lymph node > 1 cm on CT scan or hypermetabolic on FDG-PET in at least one approachable lymph nodal station for which a diagnostic cyto-histological assessment is required for clinical purpose. Patients will be randomized 1:1:1 (no suction : passive suction with EBUS dedicated syringe : manual suction with Cameco syringe) by a computer-generated random-allocation system to undergo EBUS-TBNA with one of the three different aspiration techniques. The pathologist provides a final diagnosis and, as secondary endpoint, a qualitative assessment of the sample quality using both a binary and a semi-quantitative score.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18years;
* presence of at least one hilar/mediastinal adenopathy >1 cm on short axis assessed by contrast-enhanced CT scan and/or hypermetabolic adenopathy assessed by FDG-PET;
* ability to give an informed consent

Exclusion Criteria:

* coagulopathy or bleeding diathesis that cannot be corrected;
* severe refractory hypoxemia;
* unstable hemodynamic status;
* inability to give an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-06-26 (Estimated); Study Completion 2024-06-26 (Estimated)

PRIMARY OUTCOMES:
To compare the diagnostic yield of active suction vs passive suction vs no suction EBUS-TBNA in the diagnosis of hilar/mediastinal adenopathies | 36 months
  The diagnostic yield is defined as the rate of diagnoses/total of cases. Assuming that the best technique provides a diagnostic yield of 94%, the non inferiority is defined if the difference between the best and the worst method is less than 3% with a non-inferiority limit of 10%.

SECONDARY OUTCOMES:
Adeguacy for molecular assessment in lung cancer | 36 months
  Considering only the lung cancer diagnoses, the sample is considered adeguated is if provides all the available molecular evaluations included PD-L1 iperexpression
Qualitative evaluation of the sample by the pathologist | 36 months
  The sample is evaluated by a pathologist that provides a semi-quantitative assessment of the sample, through a cell count: the sample is adeguate only if it contains more than diagnostic 100 cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Diseases Unit, Department of Immunoallergic and Respiratory Diseases, Azienda Ospedaliero Universitaria 'Ospedali Riuniti' Ancona, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Labarca G, Folch E, Jantz M, Mehta HJ, Majid A, Fernandez-Bussy S. Adequacy of Samples Obtained by Endobronchial Ultrasound with Transbronchial Needle Aspiration for Molecular Analysis in Patients with Non-Small Cell Lung Cancer. Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2018 Oct;15(10):1205-1216. doi: 10.1513/AnnalsATS.201801-045OC. PMID 30011388
- [Result] Wahidi MM, Herth F, Yasufuku K, Shepherd RW, Yarmus L, Chawla M, Lamb C, Casey KR, Patel S, Silvestri GA, Feller-Kopman DJ. Technical Aspects of Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration: CHEST Guideline and Expert Panel Report. Chest. 2016 Mar;149(3):816-35. doi: 10.1378/chest.15-1216. Epub 2016 Jan 12. PMID 26402427
- [Result] He X, Wu Y, Wang H, Yu G, Xu B, Jia N, Yao Z. Slow-pull capillary technique versus suction technique in endobronchial ultrasound-guided transbronchial needle aspiration for diagnosing diseases involving hilar and mediastinal lymph node enlargement. Ther Adv Respir Dis. 2020 Jan-Dec;14:1753466620907037. doi: 10.1177/1753466620907037. PMID 32103709
- [Result] Lin X, Ye M, Li Y, Ren J, Lou Q, Li Y, Jin X, Wang KP, Chen C. Randomized controlled trial to evaluate the utility of suction and inner-stylet of EBUS-TBNA for mediastinal and hilar lymphadenopathy. BMC Pulm Med. 2018 Dec 7;18(1):192. doi: 10.1186/s12890-018-0751-0. PMID 30526587